CLINICAL TRIAL: NCT05678725
Title: Comparison of Transcranial Direct Current Stimulation and Transcranial Alternating Current Stimulation Treatments in Improving the Motor Performance in Parkinson's Disease
Brief Title: Transcranial Direct/ Alternating Current Stimulation for Parkinson's Disease Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anhui Medical University (Other)
Responsible Party: Principal Investigator, Junjie Bu, Associate Professor, Anhui Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: tAtDComparePD
Record Dates: First submitted 2022-12-14; First posted 2023-01-10 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-02

CONDITIONS: tACS; tDCS
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Transcranial Alternating Current Stimulation (Active Comparator): the alternating current stimulation lasted 20 mins and was delivered at 2mA (peak to peak) at 20Hz during the Simple Reaction Task(SRT), targeting the primary motor cortex. EEG should be acquired before and after the stimulation session.
  Interventions: Device: tACS
- Transcranial Direct Current Stimulation (Active Comparator): the direct current stimulation lasted 20 minutes and was delivered at 2mA during the SRT, targeting at the primary motor cortex. EEG should be acquired before and after the stimulation session.
  Interventions: Device: tDCS
- Sham Group with No Actual Stimulation (Sham Comparator): the procedure of this protocol lasted 20 minutes and was delivered at 0mA during the SRT. EEG should be acquired before and after the stimulation session.
  Interventions: Device: sham

INTERVENTIONS:
Device: tACS — used round electrodes（area:3.14cm2） and the montage of a bifrontal setup with C3 as the stimulation electrode, while the return electrode placed on the right shoulder . The dose was at 2mA, 20Hz for 20 minutes.
  Arms: Transcranial Alternating Current Stimulation
Device: tDCS — used round electrodes（area:3.14cm2） and the montage of a bifrontal setup with C3 as stimulation and C4 as return electrodes. The dose was at 2mA for 20 minutes.
  Arms: Transcranial Direct Current Stimulation
Device: sham — used round electrodes（area:3.14cm2） and the montage of a bifrontal setup with C3 as stimulation and C4 as return electrodes. The stimulation lasted for 20 minutes and included a 10-second ramp-up and 10-second ramp-down.
  Arms: Sham Group with No Actual Stimulation

SUMMARY:
To investigate the difference in the treatment efficacy between transcranial direct current stimulation and transcranial alternating current stimulation on Parkinson's disease, including the improvements in the motor, cognitive, and underlying neural mechanisms behind differences in efficacy by electroencephalography (EEG).

DETAILED DESCRIPTION:
All patients underwent a medical evaluation that include physical examinations and routine laboratory studies before and after stimulation sessions. Patients were randomly allocated to tACS, tDCS, and sham groups. There are about 20 patients in each group. Allocation was by computer generating random numbers. The decision to enroll a patient was always made prior to randomization. Patients were studied using a double-blind design. Study participants, clinical raters, and all personnel responsible for the clinical care of the patient remained masked to allocated conditions and allocation parameters. Only stimulation administrators had access to the randomization list; they had minimal contact with the patients, and no role in assessing the UPDRS(Unified Parkinson´s Disease Rating Scale), Hoehn & Yahr, and MoCA(Montreal Cognitive Assessment). Each patient would be treated for 20 minutes of transcranial electrical stimulation.

Before the stimulation session, UPDRS, Hoehn & Yahr, and MoCA were obtained by a trained investigator to assess the baseline severity of symptoms. The patients received electroencephalography (EEG) recorded during resting state for 5 minutes.

During the stimulation session, patients were asked to perform simple reaction tasks at the same time.

After the stimulation session, UPDRS, Hoehn & Yahr, and MoCA were obtained, as well as the Global Index of Safety（tES side effects） to assess adverse events of the treatment. The patients also received a measure of electroencephalography (EEG) recorded during the resting state.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of idiopathic PD according to the movement disorder society criteria
* right-handed
* no clinically known hearing or vision impairment
* no history of epilepsy, dementia, other brain disorders apart from PD, severe internal organs disease, age-related frailty, etc.

Exclusion Criteria:

* parkinsonism due to drugs, Cerebrovascular disease, encephalitis, poisoning, traumatic brain injury, etc.
* Metal implants in the head (i.e., deep brain stimulator or aneurysm clips)
* severe somatic or psychiatric disorders that require medication or routinely monitoring
* participated in other interventional studies within the past 3 months

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
the changes in UPDRS III | pre-stimulation; post-stimulation (immediate after stimulation）
  Unified Parkinson´s Disease Rating Scale Section III-motor is the sum of 18 items, each item contains 0-4 ratings, where 0=normal, 1= slight, 2= mild, 3=moderate, 4=severe.
the changes in EEG power | pre-stimulation; post-stimulation (immediate after stimulation)
  EEG recording by 8 channels EEG device.

SECONDARY OUTCOMES:
simple reaction task | pre-stimulation; post-stimulation (immediately after stimulation)
  First , there was a fixation sign"+" appearing on the screen for 0.5 s, then, after 2-5 seconds, a black dot would appear. Participants were instructed to press the space bar as fast as possible when the black dot appears in the center of the screen, to measure simple perception and sustained alertness. The changes in accuracy(ACC), reaction time(RT), and ACC/RT were calculated.
the changes in MoCA | pre-stimulation; post-stimulation (immediately after stimulation)
  Montreal Cognitive Assessment is a 30-question test to assess cognitive function.

CONTACTS AND LOCATIONS:
Overall Officials: Junjie Bu, Professor, Study Chair — Anhui Medical University
Locations (1):
- Anhui Medical University, Hefei, Anhui, China

REFERENCES:
- [Derived] Liu J, Zhu Y, Chen B, Meng Q, Hu P, Chen X, Bu J. Common and specific effects in brain oscillations and motor symptoms of tDCS and tACS in Parkinson's disease. Cell Rep Med. 2025 Apr 15;6(4):102044. doi: 10.1016/j.xcrm.2025.102044. Epub 2025 Mar 27. PMID 40154492